CLINICAL TRIAL: NCT05611944
Title: Laparotomy Wound Care With Irrigation and Negative Pressure Technique in High-risk Cases of Surgical Site Infection(SSI)-A Randomized Controlled Trial
Brief Title: Irrigation and Suction Trial to Prevent SSI
Acronym: I&S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Shazia Saaqib, Assistant Professor, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 215/RC/KEMU
Record Dates: First submitted 2022-10-29; First posted 2022-11-10 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Surgical Site Infection; Diabete Mellitus; Abdominal Hysterectomy
Keywords: suction,; Wound healing; pain; Hysterectomy
MeSH Terms: conditions — Surgical Wound Infection; Diabetes Mellitus; Pain | interventions — Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: The participants will be randomized by the random number container method into an equal number of I&S groups and control groups through the parallel assignment.
Who Masked: Outcomes Assessor
Masking Description: The groups will be masked to the Outcome assessor by assigning groups A and B instead of group names and the assessor will be kept blinded about which group is the I&S group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I&S arm (Experimental): The 150 participants of the experimental arm will be assigned to the I&S group and they will be inserted bilateral Nelton drains of 24 sizes in the subcutaneous space after the closure of the rectus sheath. Their wound will be irrigated with 500cc Normal saline at running speed followed by suction for a full day. The procedure will be repeated for three consecutive days. The drains will be removed on the fourth postoperative day.
  Interventions: Device: Irrigation and suction through subcutaneus drains
- control (No Intervention): The 150 participants of the non-intervention group will be assigned to the control arm, The wound will be closed by interrupted mattress stitches without the insertion of subcutaneous drains.

INTERVENTIONS:
Device: Irrigation and suction through subcutaneus drains — Irrigation of wound will done by attaching 500cc saline to the drain on one side and let it flow freely from the other drain followed by suction of wound by attaching 60cc suction syringes on both sides creating suction pressure for 100 cc fluid.
  Arms: I&S arm

SUMMARY:
The study will be conducted on women with risk factors for SSI assigned to gynecological surgery with an open abdominal approach. The participants will be designated to either Irrigation and suction arm by bilateral drain insertion or the control arm by randomization through the parallel assignment. The participants will be followed for the outcome for four days in the hospital and then at 4 weeks, 8 weeks and 12 weeks postoperatively. The primary outcome measure will be the SSI rate. Secondary outcomes will be signs of SSI, post-operative pain, other complications and patient satisfaction.

DETAILED DESCRIPTION:
This study will be carried out in Lady willingdon Hospital, Lahore. In this study, we will recruit middle-aged and elderly diabetic women who have been assigned to open abdominal hysterectomy due to different gynaecological reasons. This cohort is at great risk of surgical site infection and other risk factors of SSI like hypertension, hepatitis and malignancy may coexist in these women. The study period will span to include three hundred participants as calculated according to sample size. The women will be divided into either an I&S group or a control group by a simple random number container method. The women in the I&S group will be inserted with bilateral drains during surgery in subcutaneous tissue after the closure of the rectus sheath and irrigated with saline followed by suction through syringe suction attached to the wound for rest of the day. The procedure will continue for three days. On the fourth day, drains are removed and stitches are removed on the fourth postoperative day. In the control group, the wound will be closed by interrupted stitches without the insertion of subcutaneous drains. The dressing will be done daily for seven days. patients with no symptoms and signs of SS will be sent home on the eighth postoperative day. The patients will be followed for symptoms of SSI, pain, readmission rate, and other complications at 4,8 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* age above 40years
* BMI>25kg/m2
* assigned to hysterectomy
* fit for anaesthesia
* patients with other medical disorders like hepatitis and hypertension will also be included in the study.

Exclusion Criteria:

* a BMI of less than 25kg/m2
* a preoperative haemoglobin level of less than 10 g/dl.

Ages: 41 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
SSI rate | first postoperative day to eighth postoperative day
  number(proportion)of surgical site infections in Intervention and control group

SECONDARY OUTCOMES:
length of wound disruption | at the time of diagnosis
  proportion of wound involved
Depth of wound disruption | at the time of diagnosis
  involving skin margins=1,subctaneous tissue=2,rectus sheath=3,peritoneum=4, 4 is the worst outcome
pain score during hospital stay | from first postoperative day to eightth postoperative day
  composit mean pain score from 0-10, 10 will be maximum adverse outcome
pain score after discharge | from discharge to completion of 12 postoperative weeks
  composite mean pain scorefrom 0-10, 10 will be maximum adverse outcome on week4, week8, week12
Other complications | from discharge to completion of 12 postoperative weeks
  complications of wound in I&S group and control group
patient satisfaction | at12th postoperative weeks completion
  not satisfied=0, satisfied=1,very satisfied=2,2 is best outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mohammmad Khalid, MBBS,MHM, Study Director — Pakistan Institute of Cardiology
Locations (1):
- Lady Willingdon Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The IPD will be shared after publication of the study.

REFERENCES:
- [Background] Flow Investigators. Fluid lavage of open wounds (FLOW): design and rationale for a large, multicenter collaborative 2 x 3 factorial trial of irrigating pressures and solutions in patients with open fractures. BMC Musculoskelet Disord. 2010 May 6;11:85. doi: 10.1186/1471-2474-11-85. PMID 20459600
- [Result] Hasan MY, Teo R, Nather A. Negative-pressure wound therapy for management of diabetic foot wounds: a review of the mechanism of action, clinical applications, and recent developments. Diabet Foot Ankle. 2015 Jul 1;6:27618. doi: 10.3402/dfa.v6.27618. eCollection 2015. PMID 26140663
- [Result] Ivanzov S, Soynov I, Kulyabin Y, Zubritskiy A, Voitov A, Omelchenko A, Arkhipov A, Bogachev-Prokophiev A. Vacuum-assisted closure versus closed irrigation for deep sternal wound infection treatment in infants: a propensity score-matched study. Interact Cardiovasc Thorac Surg. 2019 Nov 1;29(5):776-782. doi: 10.1093/icvts/ivz167. PMID 31361302